CLINICAL TRIAL: NCT06093269
Title: Pharmacokinetics Study of Cefazolin in Hemodialysis (CEFAZODIAL)
Acronym: CEFAZODIAL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR220268; EuCT number (Other: 2023-506734-73-00)
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis Catheter Infection; Infection, Bacterial
Keywords: Cefazolin; Pharmacology; Nephrology; Hemodialysis; Infectiology
MeSH Terms: conditions — Bacterial Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefazolin (Experimental): 20mg/kg to be administered in the hemodialysis circuit at the end of the 4-hour dialysis period, with no dosage adjustment planned afterwards.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — For all subjects (short kinetics):
  * Pre-injection of cefazolin
  * Start of next dialysis
  * Two hours after start of subsequent dialysis
  * End of next dialysis, before cefazolin administration
  Only in hospitalized subjects (rich kinetics):
  * 30 minutes, 1h and 2h after cefazolin injection, to describe the cefazolin peak and possible post-dialysis rebound
  * 12h, 24h and 36h after cefazolin injection, to better describe cefazolin elimination and distribution

SUMMARY:
In chronic hemodialysis patients, bacteremia is most commonly caused by dialysis catheter infections. It is estimated that the vast majority (52-84%) of these infections are due to Gram-positive cocci, particularly Staphylococcus aureus (21-43%). Penicillin M (oxacillin and cloxacillin in France) is the reference beta-lactam for the treatment of invasive methicillin-sensitive S. aureus (MSSA) infections, but has not shown a prognostic benefit in large retrospective cohorts comparing penicillin M and cefazolin, at the expense of more frequent adverse events. Dosage in the chronic hemodialysis population is unclear because it is based on old studies.

DETAILED DESCRIPTION:
In chronic hemodialysis patients, bacteremia is most commonly caused by dialysis catheter infections. It is estimated that the vast majority (52-84%) of these infections are due to Gram-positive cocci, particularly Staphylococcus aureus (21-43%). The uremia associated with kidney replacement therapy affects the immune system as a whole and is associated with an increased risk of infection. Bacterial infections are a major cause of mortality and morbidity in these patients. They are a major cause of hospitalization and the third leading cause of death after cardiovascular disease and treatment discontinuation.

Penicillin M (oxacillin and cloxacillin in France) is the reference beta-lactam for the treatment of invasive methicillin-sensitive S. aureus (MSSA) infections, but large retrospective cohorts comparing penicillin M and cefazolin have shown no prognostic benefit at the expense of more frequent adverse events. What's more, its short half-life means that it requires a more time-consuming hemodialysis protocol. Cefazolin is therefore the preferred treatment for invasive MSSA infections in the target population. This is because its clearance is slow in chronic renal failure patients during the replacement phase, and it can be administered as a single dose during hemodialysis sessions. The most recent French recommendations for cefazolin plasma concentration targets are to maintain the free form concentration at more than 4 times the minimum inhibitory concentration (MIC) for documented invasive MSSA infections or 40 - 80 mg/L (total form) for probabilistic treatment.

However, the pharmacokinetics of cefazolin at these high doses have been little studied in renal failure and dialysis patients, and dosing recommendations are mainly based on the doses recommended in the Summary of Product Characteristics (500mg at each hemodialysis session) up to 2-3g according to later pharmacokinetic and efficacy studies, or a fairly similar dosage but adapted to the weight of each patient (20mg/kg).

To our knowledge, there are no pharmacokinetic studies in infected chronic hemodialysis patients using modern assessment tools. Given the high interest in this drug in the target population, it seems essential to conduct such a study. In a second phase, a larger study could be conducted to validate the doses proposed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 or over
2. On chronic intermittent dialysis
3. With a stated indication for initiation of cefazolin either:

   1. For probabilistic treatment of a clinical presentation suggestive of MSSA infection
   2. for treatment of Gram-positive cocci bacteremia
4. With the possibility of taking peripheral blood samples or samples from the dialysis machine until the next dialysis session at 48 hours.
5. Included within a maximum of one week after the first cefazolin injection.
6. Affiliated with French social security
7. Having signed an informed consent form

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Dialysis lasting less than 3 hours, which most often corresponds to "acute" dialysis or the start of chronic dialysis, which fundamentally changes the elimination profile.
3. Allergy to cephalosporin and penicillin antibiotics (5-10% risk of cross-reactivity).
4. Non-anuric subjects with inhibitors of tubular creatinine secretion:

   1. Curative-dose trimethoprim
   2. Cimetidine
   3. Ritonavir, Rilpivirine, Dolutegravir, Cobicistat
5. Subjects under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time during which cefazolin plasma concentration exceeds the target concentration of 40 mg/L. | 48 hours after injection

SECONDARY OUTCOMES:
Occurrence of adverse events | Within 6 weeks of last dose
Early clinical efficacy - Persistence of fever >38°C | At 1 week from start of treatment
  Early clinical efficacy (at 1 week from start of treatment) in cefazolin-susceptible patients, defined as absence of failure, composite endpoint including:
  1. Persistence of fever >38°C
  2. Persistence of positive blood cultures for the same germ(s)
  3. Death for infectious reasons
  4. Change of antibiotic therapy due to ineffectiveness
Early clinical efficacy - Persistence of positive blood cultures for the same germ(s) | At 1 week from start of treatment
  Early clinical efficacy (at 1 week from start of treatment) in cefazolin-susceptible patients, defined as absence of failure, composite endpoint including:
  1. Persistence of fever >38°C
  2. Persistence of positive blood cultures for the same germ(s)
  3. Death for infectious reasons
  4. Change of antibiotic therapy due to ineffectiveness
Early clinical efficacy - Death for infectious reasons | At 1 week from start of treatment
  Early clinical efficacy (at 1 week from start of treatment) in cefazolin-susceptible patients, defined as absence of failure, composite endpoint including:
  1. Persistence of fever >38°C
  2. Persistence of positive blood cultures for the same germ(s)
  3. Death for infectious reasons
  4. Change of antibiotic therapy due to ineffectiveness
Early clinical efficacy - Change of antibiotic therapy due to ineffectiveness | At 1 week from start of treatment
  Early clinical efficacy (at 1 week from start of treatment) in cefazolin-susceptible patients, defined as absence of failure, composite endpoint including:
  1. Persistence of fever >38°C
  2. Persistence of positive blood cultures for the same germ(s)
  3. Death for infectious reasons
  4. Change of antibiotic therapy due to ineffectiveness
Late clinical efficacy - Persistence of positive blood cultures | At 6 weeks from the start of treatment
  Late clinical efficacy (at 6 weeks from the start of treatment) in patients with cefazolin-susceptible organisms, defined as absence of failure, composite endpoint including :
  1. Persistence of positive blood cultures
  2. Recurrence of initial infection
  3. Infectious death
  4. Change of antibiotic therapy due to ineffectiveness
Late clinical efficacy - Recurrence of initial infection | At 6 weeks from the start of treatment
  Late clinical efficacy (at 6 weeks from the start of treatment) in patients with cefazolin-susceptible organisms, defined as absence of failure, composite endpoint including :
  1. Persistence of positive blood cultures
  2. Recurrence of initial infection
  3. Infectious death
  4. Change of antibiotic therapy due to ineffectiveness
Late clinical efficacy - Infectious death | At 6 weeks from the start of treatment
  Late clinical efficacy (at 6 weeks from the start of treatment) in patients with cefazolin-susceptible organisms, defined as absence of failure, composite endpoint including :
  1. Persistence of positive blood cultures
  2. Recurrence of initial infection
  3. Infectious death
  4. Change of antibiotic therapy due to ineffectiveness
Late clinical efficacy - Change of antibiotic therapy due to ineffectiveness | At 6 weeks from the start of treatment
  Late clinical efficacy (at 6 weeks from the start of treatment) in patients with cefazolin-susceptible organisms, defined as absence of failure, composite endpoint including :
  1. Persistence of positive blood cultures
  2. Recurrence of initial infection
  3. Infectious death
  4. Change of antibiotic therapy due to ineffectiveness
Persistence of fever >38°C | At 1 week from start of treatment
  All components of the composite endpoint "Early clinical efficacy" will be assessed separately.
Persistence of positive blood cultures for the same germ(s) | At 1 week from start of treatment
  All components of the composite endpoint "Early clinical efficacy" will be assessed separately.
Death for infectious reasons | At 1 week from start of treatment
  All components of the composite endpoint "Early clinical efficacy" will be assessed separately.
Change of antibiotic therapy due to ineffectiveness | At 1 week from start of treatment
  All components of the composite endpoint "Early clinical efficacy" will be assessed separately.
Persistence of positive blood cultures | At 6 weeks from the start of treatment
  All components of the composite endpoint "Late clinical efficacy" will be assessed separately.
Recurrence of initial infection | At 6 weeks from the start of treatment
  All components of the composite endpoint "Late clinical efficacy" will be assessed separately.
Infectious death | At 6 weeks from the start of treatment
  All components of the composite endpoint "Late clinical efficacy" will be assessed separately.
Change of antibiotic therapy due to ineffectiveness | At 6 weeks from the start of treatment
  All components of the composite endpoint "Late clinical efficacy" will be assessed separately.
Characterizing the pharmacokinetic variability of Cefazolin | 48 hours after injection
  Characterizing the pharmacokinetic variability of Cefazolin with the occurrence of under- or over-exposure (concentration below 40 mg/L or above 80mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin MAISONS, MD, Study Director — University Hospital, Tours; Adrien LEMAIGNEN, MD-PhD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Department of hemodialysis, University Hospital of Tours, Orléans
  - Department of hemodialysis, University Hospital of Tours, Tours